CLINICAL TRIAL: NCT02321943
Title: Anomalous Self-Experience in First Episode Psychosis - A Six-Year Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 150281
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Affective Disorders, Psychotic; Self Concept
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Affective Disorders, Psychotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests including cardiovascular risk factors and immunological parameters (cytokines).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Follow-Up Group: An earlier investigated cohort with first episode psychosis patients from two Norwegian counties. Being between 18 - 65 years old and being consecutive in- or outpatient referred to first adequate treatment for a DSM-IV diagnosis of schizophrenia, bipolar disorder, or "other psychosis".

SUMMARY:
The objective of this study is to explore the longitudinal course of self-disturbances (SD) in schizophrenia. The main aim of the study is to investigate, in a 6-7-year follow-up of a representative sample of patients with first-episode schizophrenia, bipolar disorder and other psychoses. The overall aim is to expand our knowledge about the role of SDs in psychotic disorders. Increased knowledge here will aid diagnosis and treatment. The current study is a seven year follow-up of this representative cohort, with baseline measures of SDs and a comprehensive clinical and neurocognitive assessment battery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated and completed base-line part of the study,
* Patients with concurrent substance use disorder are included, but have to demonstrate at least one month without substance use, or clear signs that the psychotic disorder had started before the onset of significant substance use.

Exclusion Criteria:

* Patients with brain injury,
* Patients with on going substance use,
* Unable to provide informed consent statement.
* Not able to be interviewed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reffered to their first adequate treatment for broadly defines psychotic disorders (inkluding both schizophrenia - and bipolar Spectrum disorders) in Oppland and Hedmark counties in Norway, in 2008 - 2009 participated the base-line part of the study(E. Haug, 2012).
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in EASE (Examination of Anomalous Self-Experience)Total Score and Subscales of EASE | 6 year

SECONDARY OUTCOMES:
Change from Baseline for Structured Clinical Interview for the DSM ( SCID-I)(DSM-IV) | 6 year

OTHER OUTCOMES:
Change From Baseline in Positive and negative syndrome | 6 year
  Positive and Negative Syndrome Scale (PANSS) Total Score and Subscales of PANSS
Change From Baseline in Calgary Depression Scale Score for Schizophrenia (CDSS) | 6 year
Change from Baseline for Alcohol and Drug Use Disorder Identification Test (AUDIT and DUDIT) | 6 year
Change from Baseline for neurocognitive tests battery | 6 year
Change from Baseline for Global Assessment of Functioning - split Version(GAF) | 6 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sykehuset Innlandet HF, Brumunddal, Norway

REFERENCES:
- [Background] Haug E, Oie M, Andreassen OA, Bratlien U, Nelson B, Aas M, Moller P, Melle I. Anomalous self-experience and childhood trauma in first-episode schizophrenia. Compr Psychiatry. 2015 Jan;56:35-41. doi: 10.1016/j.comppsych.2014.10.005. Epub 2014 Oct 16. PMID 25458477
- [Background] Haug E, Oie M, Andreassen OA, Bratlien U, Raballo A, Nelson B, Moller P, Melle I. Anomalous self-experiences contribute independently to social dysfunction in the early phases of schizophrenia and psychotic bipolar disorder. Compr Psychiatry. 2014 Apr;55(3):475-82. doi: 10.1016/j.comppsych.2013.11.010. Epub 2013 Nov 28. PMID 24378241
- [Background] Haug E, Lien L, Raballo A, Bratlien U, Oie M, Andreassen OA, Melle I, Moller P. Selective aggregation of self-disorders in first-treatment DSM-IV schizophrenia spectrum disorders. J Nerv Ment Dis. 2012 Jul;200(7):632-6. doi: 10.1097/NMD.0b013e31825bfd6f. PMID 22759943
- [Background] Haug E, Oie M, Melle I, Andreassen OA, Raballo A, Bratlien U, Lien L, Moller P. The association between self-disorders and neurocognitive dysfunction in schizophrenia. Schizophr Res. 2012 Mar;135(1-3):79-83. doi: 10.1016/j.schres.2011.11.015. Epub 2011 Dec 3. PMID 22137461
- [Background] Haug E, Melle I, Andreassen OA, Raballo A, Bratlien U, Oie M, Lien L, Moller P. The association between anomalous self-experience and suicidality in first-episode schizophrenia seems mediated by depression. Compr Psychiatry. 2012 Jul;53(5):456-60. doi: 10.1016/j.comppsych.2011.07.005. Epub 2011 Aug 25. PMID 21871617